CLINICAL TRIAL: NCT03450772
Title: Open-label, Multicenter, Randomized, Cross-Over, Equivalence Study to Compare the Efficacy and Safety of Two Strengths of Pancreatin Enteric-Coated Capsules in Pancreatic Exocrine Insufficiency in Chinese Subjects
Brief Title: Equivalence Study to Compare Two Strengths of Creon in China
Acronym: CREON
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PANC3016
Record Dates: First submitted 2018-02-15; First posted 2018-03-01 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Pancreatic Insufficiency
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Creon® 25000 then Creon® 10000 (Experimental): Pancreatic enzyme
  Interventions: Drug: Creon® 25000
- Creon® 10000 then Creon® 25000 (Active Comparator): Pancreatic enzyme
  Interventions: Drug: Creon® 10000

INTERVENTIONS:
Drug: Creon® 25000 — Experimental drug
  Arms: Creon® 25000 then Creon® 10000
Drug: Creon® 10000 — Active comparator
  Arms: Creon® 10000 then Creon® 25000

SUMMARY:
This will be an open-label, randomized, multicenter, cross-over study in 60 subjects with PEI delivering data of 60 subjects for Pancreatin Enteric-Coated Capsules 25000 and of 60 subjects for Pancreatin Enteric-Coated Capsules 10000. The study will be conducted in up to 10 sites in China.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Subjects ≥ 18 years
* A) Chronic pancreatitis must be documented in the medical file by at least one of the following methods:

  * Imaging techniques (ultrasound, CT, MRI, or endoscopic ultrasound)
  * ERCP (endoscopic retrograde cholangiopancreatography)
  * Plain film of the abdomen with pancreatic calcification or
* B) Partial or total pancreatectomy ≥ 30 days prior to enrollment and without current postsurgery complications
* PEI proven by human fecal elastase ≤ 100 µg/g stool (during the screening period)
* Subjects without Creon (Pancreatin Enteric Coated Minimicrospheres) intake in the past three months
* Females of child-bearing potential should agree to continue using a medically acceptable method of birth control throughout the study and for 30 days immediately after the last dose of study drug. Medically acceptable methods of birth control include bilateral tubal ligation or the use of either a contraceptive implant, a contraceptive injection (e.g. Depo-Provera™), an intrauterine device, or an oral contraceptive taken within the past three months where the subject agrees to continue using during the study or to adopt another birth control method, or a double-barrier method which consists of a combination of any two of the following: diaphragm, cervical cap, condom, or spermicide

Exclusion Criteria:

* Subjects with a history of fibrosing colonopathy
* Solid organ transplant
* Surgery affecting the stomach or bowel, except pancreatectomy or appendectomy
* Surgery affecting the stomach or bowel, except pancreatectomy or appendectomy
* Subjects with recurrent malignant tumors of any kind
* Use of an immunosuppressive drug or chemotherapy
* Acute phase of pancreatitis
* Acute phase of pancreatitis
* Subjects who are not able or willing to ingest 90g fat/day (± 10 g fat/day) during the cross-over periods or are not willing to collect complete stools during the demarcation period.
* Subjects in an instable condition after pancreatic surgery (Karnofsky index < 70)
* Known infection with HIV
* Pregnancy or lactation
* Current excessive alcohol intake or drug abuse
* Investigational drug intake within prior 30 days
* Known allergy against pancreatin of porcine origin or to any of the excipients of Pancreatin Enteric-Coated Capsules
* Suspected non-compliance or non-cooperation
* Celiac disease, Crohn´s disease
* Ileus or acute abdomen in the medical history
* Mental disability or any other lack of fitness, in the investigator's opinion, to preclude subject's participation in or to complete the study
* Any acute or chronic disease (i.e infectious diseases) which may limit the hospitalization, dietary adherence or stool collection or completion of the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-08-31 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Coefficient of fat absorption | 5 days

SECONDARY OUTCOMES:
fat intake - fat excretion/fat intake x 100 | 5 days
stool weight | 5 days
Clinical symptomatology | 5 days and 24 weeks
  stool frequency, stool consistency, abdominal pain, flatulence
Subject's acceptance of treatment and preference | 5 days and 24 weeks
  Subject's acceptance of treatment will be judged based on the following scale: very good, good, moderate and unsatisfactory.
  Which treatment did you prefer? No difference between treatment 1 and treatment 2 Treatment 1 is better than treatment 2 Treatment 2 is better than treatment 1

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changhai Hospital, Shanghai, China